CLINICAL TRIAL: NCT00912379
Title: Comparison of the Hemoglobin Results Obtained With the Masimo SpHb™ Device and the Clinical Laboratory Measurement
Brief Title: Hemoglobin Measured by MASIMO SpHb™ Device and Laboratory Measurement
Status: Completed | Type: Observational
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Other Study IDs: 2009/10
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Patients' Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- hemoglobin determination: ICU and emergency unit patients
  Interventions: Biological: hemoglobin determination

INTERVENTIONS:
Biological: hemoglobin determination — laboratory and non invasive hemoglobin determinations

SUMMARY:
The purpose of this study is to compare the hemoglobin results obtained with the Masimo SpHb™ device and the Clinical Laboratory.

ELIGIBILITY:
Inclusion Criteria:

* emergency unit patients, PACU (post-anaesthesia care unit) and ICU patients requiring an hemoglobin determination

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: emergency unit patients and ICU patients requiring an hemoglobin determination
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2009-06; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Accuracy of the Masimo Labs Pulse-Hemoglobin-Meter Monitor | End of the period of recruitment

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Foch, Suresnes, France